CLINICAL TRIAL: NCT06108544
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Placebo- and Active Comparator-Controlled Study With a Randomized Withdrawal and Retreatment Period to Evaluate the Efficacy, Safety, and Tolerability of TAK-279 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study About How Well TAK-279 Works and Its Safety in Participants With Moderate-to-severe Plaque Psoriasis During 60 Weeks of Treatment With a Withdrawal and Retreatment Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-279-3002; 2023-505842-24-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Plaque Psoriasis
Keywords: Drug Therapy; Latitude Psoriasis 2, Latitude Research Program
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-279 (Experimental)
  Interventions: Drug: TAK-279
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Apremilast (Active Comparator)
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: TAK-279 — Specified drug on specified days.
  Arms: TAK-279
Drug: Placebo — Specified drug on specified days.
  Arms: Placebo
Drug: Apremilast — Specified drug on specified days.
  Arms: Apremilast

SUMMARY:
The main aim of this study is to show how well TAK-279 reduces the skin plaques compared to placebo, in participants with moderate-to-severe plaque psoriasis. Participants will be assigned to one of the 3 study treatments (TAK-279, apremilast (an approved treatment), or a placebo). Participants will be in the study for up to 69 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-279. TAK-279 is being tested to treat people with moderate to severe plaque psoriasis.

The study will enroll approximately 1000 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups for TAK-279, placebo, or apremilast in a ratio of 2:1:1 which will remain undisclosed to the patient and investigator during the study (unless there is an urgent medical need):

* TAK-279
* Apremilast
* Placebo

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 69 weeks. Participants will go through a screening process to make sure they meet the rules for taking part in the study. This will take up to 35 days. If participants meet the study rules, they will be treated for up to 60 weeks. There will be a safety follow-up visit 4 weeks after their last day of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Plaque psoriasis for at least 6 months.
2. Moderate to severe disease.
3. Candidate for phototherapy or systemic therapy.

Exclusion Criteria:

1. Other forms of psoriasis.
2. History of recent infection.
3. Prior exposure to TAK-279 or active comparator.

Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving ≥75% Improvement from Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving 90% Improvement from Baseline in PASI (PASI-90) at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. Higher scores indicate worsening. 'Clear' will include all participants who score a 0.
Percentage of Participants Achieving PASI-100 at Week 16 Comparing TAK-279 Against Placebo | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving a Scalp-specific Physician's Global Assessment (ssPGA) of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants Achieving PASI-75 at Week 4 Comparing TAK-279 Against Placebo | Week 4
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants with a Baseline Dermatology Life Quality Index (DLQI) Score ≥2 who Achieve DLQI Score of 0 or 1 at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Percentage of Participants With a Baseline Psoriasis Symptoms and Signs Diary (PSSD) ≥1 who Achieve Weekly Mean PSSD Symptom Score of 0 at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Change from Baseline in Nail Psoriasis Severity Index (NAPSI) at Week 16 Among Participants With Nail Involvement at Baseline Comparing TAK-279 Against Placebo | Baseline, Week 16
  The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lunula, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each nail will be scored for both nail matrix and nail bed psoriasis for each quadrant (ranging from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores indicate more severe psoriasis.
Change from Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16 Comparing TAK-279 Against Placebo | Week 16
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percentage Change from Baseline in BSA Affected by Psoriasis at Week 16 Comparing TAK-279 Against Placebo | Week 16
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percentage of Participants Achieving a Physician's Global Assessment (PGA) of the Hands and/or Feet of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease From Baseline at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  PGA is a 5-point scale and a score of 0 to 4 should be assigned, based on the category that best describes the severity of active psoriasis of the participant's hands and/or feet (palmoplantar), where 0=clear and 4=severe. Higher scores indicate worsening of severity. It will be evaluated for participants with the presence of active hand or foot psoriasis on Day 1.
Change from Baseline in DLQI at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life). It will be evaluated for participants with a baseline DLQI score ≥2.
Change from Baseline in the Short Form-36 Health Survey (SF-36) Version 2 Scores at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  The SF-36 is a self-administered, validated questionnaire designed to measure generic health-related QoL. This 36-item questionnaire measures 8 domains, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Two summary scores, including the physical component summary (PCS) and mental component summary (MCS), will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL.
Change from Baseline in the EuroQoL 5-Dimension 5-Level Questionnaire (EQ-5D-5L) Scores at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  EQ-5D-5L includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and 5 response levels for each domain (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). The scores in the 5 dimensions will be summarized into a health state index score. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health; 0=a health state equivalent to death, and 1=perfect health.
Change in Work Productivity and Activity Impairment-Psoriasis (WPAI-PSO) Questionnaire Scores at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work. Four scores are derived: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism and impairment in activities performed outside of work. Each WPAI score will be expressed as impairment percentages (0-100) with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Apremilast | Baseline to Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. Higher scores indicate worsening. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 24 Comparing TAK-279 Against Apremilast | Baseline to Week 24
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Change from Baseline in Weekly Mean PSSD Symptom Score at Week 16 Comparing TAK-279 Against Apremilast | Baseline to Week 16
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Percentage of Participants Achieving an ssPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Apremilast | Baseline to Week 16
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants Achieving PASI-100 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-100 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' will include all participants who score a 0.
Percentage of Participants with a Baseline DLQI Score ≥2 who Achieve DLQI Score of 0/1 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Percentage of Participants With a Baseline PSSD ≥1 who Achieve a Weekly Mean PSSD Symptom Score of 0 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Change from Baseline in NAPSI Among Participants With Nail Involvement at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lunula, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each nail will be scored for both nail matrix and nail bed psoriasis for each quadrant (ranging from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores indicate more severe psoriasis.
Percentage of Participants Achieving an ssPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 24 Comparing TAK-279 Against Apremilast | Baseline to Week 24
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Change from Baseline in DLQI at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Change from Baseline in BSA Affected by Psoriasis at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percent Change from Baseline in BSA Affected by Psoriasis at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' will include all participants who score a 0.
Percentage of Participants With a Baseline DLQI Score ≥2 who Achieve a DLQI Score of 0/1 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Percentage of Participants With a Baseline PSSD ≥1 who Achieve a Weekly Mean PSSD Symptom Score of 0 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Change from Baseline in ssPGA at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants Achieving a PGA of the Hands and/or Feet of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease From Baseline at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  PGA is a 5-point scale and a score of 0 to 4 should be assigned, based on the category that best describes the severity of active psoriasis of the participant's hands and/or feet (palmoplantar), where 0=clear and 4=severe. Higher scores indicate worsening of severity. It will be evaluated for participants with the presence of active hand or foot psoriasis on Day 1.
Change from Baseline in SF-36 Version 2 Scores at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The SF-36 is a self-administered, validated questionnaire designed to measure generic health-related QoL. This 36-item questionnaire measures 8 domains, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Two summary scores, including the PCS and MCS, will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL.
Change from Baseline in the EQ-5D-5L Scores at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  EQ-5D-5L includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and 5 response levels for each domain (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). The scores in the 5 dimensions will be summarized into a health state index score. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health; 0=a health state equivalent to death, and 1=perfect health.
Change from Baseline in the WPAI-PSO Scores at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work. Four scores are derived: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism and impairment in activities performed outside of work. Each WPAI score will be expressed as impairment percentages (0-100) with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Weeks 24 and 40 Comparing TAK-279 Against Apremilast | Baseline, Weeks 24 and 40
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Weeks 24 and 40 Comparing TAK-279 Against Apremilast | Weeks 24 and 40
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Weeks 24 and 40 Comparing TAK-279 Against Apremilast | Weeks 24 and 40
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Time to Relapse for PASI-75 Responders at Week 40 Comparing TAK-279 Against Placebo | Up to Week 60
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants With Maintenance of PASI-75 Response at Week 60 Comparing TAK-279 Against Placebo | Week 60
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants with Maintenance of sPGA of Clear (0) or Almost Clear (1) With a ≥2-Point Decrease from Baseline at Week 60 Comparing TAK-279 Against Placebo | Baseline to Week 60
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants With a Disease Relapse Comparing TAK-279 Against Placebo | Week 40
  Relapse is defined as a percent change from baseline in PASI score that is at least 50% worse than that observed at Week 40. PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Higher scores indicate worsening.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESI) | Up to week 69
  TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product. An AESI (serious or nonserious) is an adverse event of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator may be appropriate.
Number of Participants With Clinically Significant Abnormalities in Vital Signs | Up to week 69
Number of Participants With Clinically Significant Laboratory Values | Up to week 69
Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | Up to week 69

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (217):
- United States (66):
  - Total Dermatology, Birmingham, Alabama
  - Cahaba Dermatology Skin Health Center, Hoover, Alabama
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Zenith Research, Inc., Beverly Hills, California
  - UNISON Clinical Trials (Shahram Jacobs md inc.), Encino, California
  - First OC Dermatology Research Inc., Fountain Valley, California
  - Long Beach Research Institute, LLC, Long Beach, California
  - Metropolis Dermatology Downtown LA - Probity - PPDS, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - TCR Medical Corporation, San Diego, California
  - University Clinical Trials, San Diego, California
  - Dermatology Institute and Skin Care Center, Santa Monica, California
  - Revival Research Corporation - Florida - ClinEdge - PPDS, Doral, Florida
  - Florida Academic Centers Research, Miami, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - FXM Research Miramar, Miramar, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Advanced Clinical Research Institute (ACRI) - Florida, Tampa, Florida
  - Olympian Clinical Research - 6331 Memorial Hwy, Tampa, Florida
  - Divine Dermatology and Aesthetics, LLC, Atlanta, Georgia
  - Advanced Medical Research, PC, Atlanta, Georgia
  - Skin Care Physicians of Georgia, Macon, Georgia
  - NorthShore Medical Group Dermatology - Skokie, Skokie, Illinois
  - DS Research - 1005 E. Lewis & Clark Pkwy Indiana Location, Clarksville, Indiana
  - Skin Sciences, PLLC, Louisville, Kentucky
  - DS Research of Kentucky, Louisville, Kentucky
  - Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - Allcutis Research LLC, Beverly, Massachusetts
  - Beacon Clinical Research LLC, Brockton, Massachusetts
  - David Fivenson MD Dermatology PLLC, Ann Arbor, Michigan
  - University of Michigan Hospital - 1500 E Medical Center Dr, Ann Arbor, Michigan
  - Oakland Hills Dermatology - 3400 Auburn Rd, Auburn Hills, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists PC, Omaha, Nebraska
  - Vivida Dermatology - Flamingo Rd - Probity - PPDS, Las Vegas, Nevada
  - ALLCUTIS Research, LLC., Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Mount Sinai Doctors -234 E 85th St, New York, New York
  - Sadick Research Group, New York, New York
  - Derm Research Center of NY, Stony Brook, New York
  - Montefiore Dermatology - BRANY - PPDS, The Bronx, New York
  - Duke Dermatology Clinic, Durham, North Carolina
  - The Skin Surgery Center for Clinical Research - Objective Health - PPDS, Winston-Salem, North Carolina
  - Wake Forest Baptist Health Department of Dermatology - 4618 Country Club Rd, Winston-Salem, North Carolina
  - ClinOhio Research Services, Columbus, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Oregon Medical Research Center PC, Portland, Oregon
  - University of Pittsburgh Medical Center-3601 5th Ave, Pittsburgh, Pennsylvania
  - Cumberland Skin Center for Clinical Research - Objective Health - PPDS, Hermitage, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Research Center, Arlington, Texas
  - UT Physicians Dermatology - Bellaire Station, Bellaire, Texas
  - Modern Research Associates, Dallas, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - Austin Institute for Clinical Research, Inc. - Pflugerville - ClinEdge - PPDS, Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Houston Center for Clinical Research, LLC, Sugar Land, Texas
  - Center For Clinical Studies, LTD. LLP - 451 N Texas Ave, Webster, Texas
  - Center For Clinical Studies,LTD. LLP - 451 N Texas Ave, Webster, Texas
  - Virginia Clinical Research - 6160 Kempsville Cir, Norfolk, Virginia
- Argentina (5):
  - Conexa Investigación Clínica S.A., Buenos Aires
  - STAT Research S.A., Buenos Aires
  - Instituto de Neumonologia y Dermatologia, Buenos Aires
  - Centro de Investigacion Clínica - CEDIC, Ciudad Autónomade Buenos Aires
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán
- Bulgaria (16):
  - Medical Center Unimed EOOD, Sevlievo, Gabrovo
  - Medical Center Asklepii OOD, Dupnitsa, Kyustendil
  - MBAL Skin Systems, Doganovo, Elin Pelin, Sofia
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Sofia-Grad
  - Diagnostic Consultative Centre - Focus-5 - LZIP EOOD, Sofia, Sofia-Grad
  - Medical Center Hera EOOD, Sofia, Sofia-Grad
  - Diagnostic Consultative Center XXVIII - Sofia - EOOD, Sofia, Sofia-Grad
  - Ambulatory for Specialized Medical Care- Group Practice in Dermatology - Clinic EuroDerma OOD, Sofia, Sofia-Grad
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - MC Comac Medical - IRN - PPDS, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment - Dobrich AD, Dobrich
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - Diagnostic Consultative Center Sveti Georgi EOOD, Haskovo
  - Medical Center Medconsult Pleven OOD, Pleven
  - Medical Center Exacta Medica - Vasil Levski 60, Pleven
  - University Multiprofile Hospital for Active Treatment -Dr. Georgi Stranski -Gen. V. Vazov Str 91, Pleven
- Canada (22):
  - Dermatology Research Institute, Inc. - Probity - PPDS, Calgary, Alberta
  - Alberta DermaSurgery Centre - Probity - PPDS, Edmonton, Alberta
  - VIDA Dermatology - Probity - PPDS, Edmonton, Alberta
  - CaRe Clinic-Red Deer, Red Deer, Alberta
  - Wiseman Dermatology Research Inc. - Probity - PPDS, Winnipeg, Manitoba
  - Brunswick Dermatology Centre - Probity - PPDS, Fredericton, New Brunswick
  - Lima's Excellence In Allergy And Dermatology Research (Leader) Inc. - Probity - PPDS, Hamilton, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - DermEffects - Probity - PPDS, London, Ontario
  - Lynderm Research Inc - Probity - PPDS, Markham, Ontario
  - DermEdge Research - Probity - PPDS, Mississauga, Ontario
  - The Centre for Clinical Trials Inc. - Probity - PPDS, Oakville, Ontario
  - Oshawa Clinic-117 King St, Oshawa, Ontario
  - SKiN Centre for Dermatology - Peterborough - Probity - PPDS, Peterborough, Ontario
  - Centre For Dermatology and Cosmetic Surgery - Probity - PPDS, Richmond Hill, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation - Probity - PPDS, Richmond Hill, Ontario
  - Canadian Dermatology Centre - Probity - PPDS, Toronto, Ontario
  - Toronto Research Centre - Probity - PPDS, Toronto, Ontario
  - Alliance Clinical Trials - Probity - PPDS, Waterloo, Ontario
  - XLR8 Medical Research - Probity - PPDS, Windsor, Ontario
  - Siena Medical Research, Westmount, Quebec
  - Skinsense Medical Research - 411 2nd Ave N - Probity - PPDS, Saskatoon, Saskatchewan
- China (13):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital With Nanjing Medical University(Jiangsu Province Hospital), Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine - Qingchun Campus, Hangzhou, Zhejiang
  - Huashan Hospital Fudan University - PPDS, Shanghai
- Czechia (10):
  - Dermamedica, s.r.o. - Kozni Ambulance Nachod, Náchod, Královéhradecký kraj
  - Nemocnice AGEL Novy Jicin a.s, Nový Jičín, Moravskoslezský kraj
  - CCR Ostrava s.r.o., Ostrava, Moravskoslezský kraj
  - Praglandia s.r.o., Prague, Ohio
  - Dermskin s.r.o., Olomouc, Olomoucký kraj
  - CLINTRIAL s.r.o., Prague, Praha, Hlavní Mesto
  - Pratia Brno s.r.o. - PRATIA - PPDS, Brno, South Moravian
  - Pratia Pardubice a.s. - PRATIA - PPDS, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Prof. MUDr. Petr Arenberger, DrSc. - CRC - PPDS, Prague
- France (3):
  - Centre Hospitalier Le Mans, Le Mans, Ohio
  - AP-HM- Hôpital de La Timone, Marseille
  - Hôpital Charles Nicolle-1 Rue de Germont, Rouen
- Germany (7):
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Klinische Forschung Dresden GmbH (KFGN) - PRATIA - PPDS, Dresden, Saxony
  - Praxis fur Dermatologie and Venerologie, Dresden, Saxony
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - FutureMeds - Berlin - PPDS, Berlin
  - Dermatologikum Hamburg, Hamburg
  - Medizinisches Versorgungszentrum DermaKiel GmbH, Kiel
- Greece (5):
  - Hospital A.Syggros, Athens, Attica
  - University General Hospital ''ATTIKON'', Chaïdári, Attica
  - University Hospital of Ioannina, Loannina, Loannina
  - Hospital Of Skin And Venereal Diseases of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hungary (6):
  - Szegedi Tudomanyegyetem, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus, Debrecen, Hajdú-Bihar
  - Allergo-Derm Bakos Kft- Szolnok-Baross utca 20, Szolnok, Jász-Nagykun-Szolnok
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár, Somogy County
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz, Szombathely, Vas County
  - Pécsi Tudomanyegyetem - Vasvari Pal u., Pécs
- Israel (5):
  - Hadassah Medical Center- Ein Kerem - PPDS, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center Ichilov - PPDS 27004, Tel Aviv, Tel Aviv
  - HaEmek Medical Center, Afula
  - Rabin Medical Center - PPDS, Petah Tikva
- Latvia (8):
  - Adoria, Riga, Ohio
  - Smite Aija doctor practice in dermatology, venerology, Talsi, Talsu Aprinkis
  - Semigallia, Kuldīga
  - Riga 1st Hospital, Riga
  - Health Center 4, Center of Diagnostics, Riga
  - J. Kisis, Riga
  - Veseliba un estetika, Riga
  - Health Center 4, Clinic of Dermatology, Riga
- Poland (35):
  - Solumed Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Twoja Przychodnia PCM, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne ALL-MED, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne - FutureMeds - PPDS, Krakow, Lesser Poland Voivodeship
  - WroMedica, Wroclaw, Lower Silesian Voivodeship
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Dorota Krasowska, Lublin, Lublin Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne sp. z o.o, Nowa Sól, Lubusz Voivodeship
  - Centrum Terapii Wspolczesnej, Lódz, Lódzkie
  - ClinMedica Research, Skierniewice, Lódzkie
  - ETG Siedlce - PPDS, Siedlce, Masovian Voivodeship
  - RCMed Oddzial Sochaczew, Sochaczew, Masovian Voivodeship
  - Clinical Research Group Sp. z o.o, Warsaw, Masovian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - ETG Warszawa - PPDS, Warsaw, Masovian Voivodeship
  - FutureMeds - Targowek - PPDS, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Torun - MICS - PPDS, Torun, Ohio
  - NZOZ Osteo Medic SC Artur Racewicz Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Chojnice - PRATIA - PPDS, Chojnice, Pomeranian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Silesian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - Centrum Uslug Medycznych MaxMed, Bochnia
  - Ambulatorium Barbara Bazela, Elblag
  - Globe Badania Kliniczne Spólka z o.o. - Klodzko, Klodzko Dolnoslaskie
  - MCM Krakow - PRATIA - PPDS, Krakow
  - Diamond Clinic, Krakow
  - ETG Lublin - PPDS, Lublin
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - DermoDent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski, s.c., Osielsko
  - Royalderm, Warsaw
  - dermMEDICA Sp. z o.o, Wroclaw
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
  - Ostrowieckie Centrum Medyczne, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- GCM Medical Group, PSC -62 Calle Jose Marti, San Juan, Puerto Rico
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Manises, Manises, Valencia
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
- United Kingdom (9):
  - Velocity Clinical Research, High Wycombe - PPDS, High Wycombe, Buckinghamshire
  - 4 Medical Clinical Solutions (4MCS) Swinton - PPDS, Ilford, Essex
  - Accellacare of Yorkshire, Chorley, Lancashire
  - Salford Royal Hospital - PPDS, Salford, Lancashire
  - Whipps Cross Hospital, London, London, City of
  - Accellacare of Northamptonshire, Harrow, Middlesex
  - Velocity Clinical Research, North London - PPDS, London, Middlesex
  - Accellacare - North London Clinical Studies Centre, Northwood, Middlesex
  - St Luke's Hospital, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/516bd1c8c4dd4621